CLINICAL TRIAL: NCT00792792
Title: Non-contact, Intra-operative & Post-operative Device, Evaluation of Tissue Transfer Flaps After Reconstructive Surgery.
Brief Title: Monitoring of Tissue Transfer Flaps by Modulated Imaging
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial study.
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Gregory Evans, M.D., Chair, Department of Plastic Surgery, University of California, Irvine
Other Study IDs: 20075891
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Other Reconstructive Surgery
Keywords: tissue transfer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tissue transfer skin flap: Modulated Imaging Spectroscopy
  Interventions: Device: Modulated Imaging

INTERVENTIONS:
Device: Modulated Imaging — Modulated Imaging Spectroscopy

SUMMARY:
Tissue transfer flaps are a method of moving tissue from a donor location to a recipient location. In the case of a free tissue transfer flaps, the blood vessels to the transferred tissues are detached and then re-attached to different arteries and veins at the recipient site. The process of reconstructive surgery using tissue transfer flaps is not without complications. These complications may include acute arterial or venous occlusion, as well as the development of late complications such as fat necrosis and flap atrophy.

DETAILED DESCRIPTION:
The researchers developed a safe, non-contact, intra-operative and post-operative device called Modulated Imaging, can detect changes in a flap's optical properties and can correlate with arterial or venous occlusion or with the development of fat necrosis or flap atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older planned to undergo reconstructive surgery

Exclusion Criteria:

* All emergency reconstructive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from Surgical Department as outpatients and in-patient bases that require reconstructive surgery using a pedicle or free tissue transfer flap.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Transfer Skin flap | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Evans R Gregory, PhD, Principal Investigator — Aesthetic & Plastic Surgery Institute, UCIMC
Locations (1):
- University of California Medical Center, Orange, California, United States